CLINICAL TRIAL: NCT00564512
Title: Randomized Phase-III Trial Comparing Fludarabine and Cyclophosphamide Plus Rituximab (FCR) to FC and MabCampath (FCCam) for Previously Untreated Fit Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Fludarabine, Cyclophosphamide, and Rituximab or Alemtuzumab in Treating CLL2007 CLL 2007 FMP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000577580; CLL-2007-FMP (Other: GOELAMS)
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2009-04

CONDITIONS: Leukemia
Keywords: B-cell chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; Rituximab; Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FCCAM (Experimental): Fludarabine-Cyclophosphamide-Campath (FCCam) Oral Fludarabine: 40 mg/m2 per os, D1 to D3 Oral Cyclophosphamide: 250 mg/m2/day as one dose at noon, D1 to D3 Campath®: 30 mg sc, D1 to D3 without dose escalation
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: fludarabine
- FCR (Active Comparator): Fludarabine-Cyclophosphamide-Rituximab (FCR)
  First course:
  Rituximab 375 mg/m2 on D1.
  D2 to D4:
  oral Fludarabine: 40 mg/m2/day as a single morning dose oral Cyclophosphamide: 250 mg/m2/day as a single dose at noon
  Subsequent courses (2 to 6)
  Rituximab 500 mg/m2 on D1
  D1 to D3:
  oral Fludarabine: 40 mg/m2/day as a single morning dose oral Cyclophosphamide: 250 mg/m2/day as a single dose at noon
  Interventions: Biological: Campath; Drug: cyclophosphamide

INTERVENTIONS:
Biological: Campath — Fludarabine-Cyclophosphamide-Campath (FCCam)
  Other Names: Alemtuzumab
  Arms: FCR
Biological: rituximab — Fludarabine-Cyclophosphamide-Rituximab (FCR)
  Other Names: Mabthera®
  Arms: FCCAM
Drug: cyclophosphamide — Fludarabine-Cyclophosphamide-Campath (FCCAM) Fludarabine-Cyclophosphamide-Rituximab (FCR)
  Other Names: Endoxan®
Drug: fludarabine — Fludarabine-Cyclophosphamide-Campath (FCCAM) Fludarabine-Cyclophosphamide-Rituximab (FCR)
  Other Names: Fludara®
  Arms: FCCAM

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine and cyclophosphamide, work in different ways to kill cancer cells or stop them from growing. Monoclonal antibodies, such as rituximab and alemtuzumab, can block cancer growth in different ways. Some find cancer cells and help kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. It is not yet known whether giving fludarabine and cyclophosphamide together with rituximab is more effective than giving fludarabine and cyclophosphamide together with alemtuzumab in treating B-cell chronic lymphocytic leukemia.

PURPOSE: This randomized phase III trial is studying giving fludarabine together with cyclophosphamide and rituximab to see how well it works as first-line therapy compared with giving fludarabine together with cyclophosphamide and alemtuzumab in treating patients with B-cell chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare 36-month progression-free survival in patients with Binet stage B or C B-cell chronic lymphocytic leukemia treated with first-line therapy comprising fludarabine phosphate and cyclophosphamide and either rituximab or alemtuzumab.

Secondary

* To compare the disease-free survival, event-free survival, and overall survival of patients treated with these regimens.
* To compare time to next treatment in patients treated with these regimens.
* To compare the overall response rate (complete response [CR] and partial response [PR]) in patients treated with these regimens.
* To compare the rate of phenotypic and molecular response in patients treated with these regimens.
* To compare the duration of phenotypic, molecular, complete and partial responses in patients treated with these regimens.
* To compare the response rates and survival times in biological subgroups.
* To compare the rates of treatment-related adverse effects in patients treated with these regimens.
* To compare the quality of life of patients treated with these regimens.
* Minimal residual disease study.

OUTLINE: This is a multicenter study. Patients are stratified according to Ig mutational status and cytogenetic abnormalities. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive rituximab IV on day 1 and fludarabine phosphate and cyclophosphamide IV or orally on days 2-4 of course 1. Beginning in course 2 and for all subsequent courses, patients receive rituximab IV on day 1 and fludarabine phosphate and cyclophosphamide IV or orally on days 1-3.
* Arm II: Patients receive alemtuzumab subcutaneously, oral fludarabine phosphate, and oral cyclophosphamide on days 1-3.

In both arms, treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion

Diagnosis of B-cell chronic lymphocytic leukemia (CLL), meeting the following criteria:

* Binet classification stages B or C
* Del 17 p (FISH) negative (< 10 % positives cores)
* Matutes score 4 or 5

Exclusion Transformation to aggressive B-cell malignancy (e.g. diffuse large cell lymphoma, Hodgkin lymphoma, or prolymphocytic leukemia)

PATIENT CHARACTERISTICS:

Exclusion ECOG performance status ≥ 2

* Life expectancy < 6 months
* Creatinine clearance < 60 mL/min
* Total bilirubin > 2 x upper limit of normal (ULN)
* Gamma glutamyltransferase or transaminase levels > 2 x ULN
* Cumulative illness rating scale > 6
* HIV seropositivity
* Hepatitis B or C seropositivity (unless clearly due to vaccination)
* Clinically significant autoimmune anemia
* Active bacterial, viral, or fungal infection
* Active second malignancy currently requiring treatment (except basal cell carcinoma or in situ endometrial carcinoma) and/or less than 5 years complete remission after breast cancer
* Any severe comorbid conditions including, but not limited to, any of the following:

  * Class III or IV heart failure
  * Recent myocardial infarction
  * Unstable angina
  * Ventricular tachyarrhythmias requiring ongoing treatment
  * Severe chronic obstructive pulmonary disease with hypoxemia
  * Uncontrolled diabetes mellitus
  * Uncontrolled hypertension
* Concomitant disease requiring prolonged use of corticosteroids (> 1 month)
* Known hypersensitivity with anaphylactic reaction to humanized monoclonal antibodies or any of the study drugs
* Contraindication to the use of rituximab or alemtuzumab according to Summary of Product Characteristics
* Any coexisting medical or psychological condition that would preclude participation in the required study procedures
* Any mental deficiency preventing proper understanding of the requirements of treatment
* Person under law control
* Pregnant or breastfeeding women
* Fertile patients who cannot or do not wish to use an effective method of contraception, during and for 12 months after the final treatment used for the purposes of the study

PRIOR CONCURRENT THERAPY:

Inclusion

* No prior chemotherapy, radiotherapy, or immunotherapy for CLL
* Corticosteroids within the past month allowed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 36 months | 36 months follow up

SECONDARY OUTCOMES:
Disease-free survival | 36 months follow up
Event-free survival | 36 months follow up
Overall survival | 36 months follow up
Time to next treatment | 36 months follow up
Overall response rate (complete response [CR] and partial response [PR]) | 36 months follow up
Duration of phenotypic, molecular, NCI complete and partial responses | 36 months follow up
Response rates and survival times in biological subgroups | 36 months follow up
Treatment-related adverse effects | 36 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Lepretre, MD, Study Chair — Centre Henri Becquerel; Pierre Feugier, Principal Investigator — CHU de Nancy - Hopitaux de Brabois; Roselyne DELEPINE, mrs, Study Director — Groupe Est Ouest Etudes leucemies et Autres Maladies du Sang
Locations (1):
- Centre Henri Becquerel, Rouen, France

REFERENCES:
- [Derived] Grgurevic S, Montilla-Perez P, Bradbury A, Gilhodes J, Queille S, Pelofy S, Bancaud A, Filleron T, Ysebaert L, Recher C, Laurent G, Fournie JJ, Cazaux C, Quillet-Mary A, Hoffmann JS. DNA polymerase nu gene expression influences fludarabine resistance in chronic lymphocytic leukemia independently of p53 status. Haematologica. 2018 Jun;103(6):1038-1046. doi: 10.3324/haematol.2017.174243. Epub 2018 Mar 22. PMID 29567785
- [Derived] Lepretre S, Aurran T, Mahe B, Cazin B, Tournilhac O, Maisonneuve H, Casasnovas O, Delmer A, Leblond V, Royer B, Corront B, Chevret S, Delepine R, Vaudaux S, Van Den Neste E, Bene MC, Letestu R, Cymbalista F, Feugier P. Excess mortality after treatment with fludarabine and cyclophosphamide in combination with alemtuzumab in previously untreated patients with chronic lymphocytic leukemia in a randomized phase 3 trial. Blood. 2012 May 31;119(22):5104-10. doi: 10.1182/blood-2011-07-365437. Epub 2012 Feb 14. PMID 22337714